CLINICAL TRIAL: NCT06664450
Title: Exploring Brain Fog Symptoms in Patients With Obstructive Sleep Apnea and CPAP Therapy Impact: A Pilot Study
Brief Title: Brain Fog in Sleep Apnea
Acronym: BF -OSA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Eleonora Volpato, Clinical Professor, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: BF-OSA
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea (OSA); Brain Fog; Cognitive Impairment; CPAP Therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Mental Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with severe OSA treated with CPAP for at least 3 months.: The group consists of patients diagnosed with severe Obstructive Sleep Apnea (OSA) who have been treated with Continuous Positive Airway Pressure (CPAP) therapy for a minimum of 3 months.
- Patients with severe OSA in new access and therefore not yet subjected to CPAP treatment.: This group comprises patients recently diagnosed with severe Obstructive Sleep Apnea (OSA) who have not yet started treatment with Continuous Positive Airway Pressure (CPAP). This cohort will be compared to a group of patients who have been undergoing CPAP therapy for at least 3 months. The primary objective is to assess the presence and severity of cognitive symptoms, commonly referred to as "Brain Fog," which includes impairments in memory, attention, and concentration. Participants in this group will complete a one-time assessment, which will involve various scales to evaluate cognitive function, sleep quality, daytime sleepiness, and fatigue levels. This study aims to provide insights into the cognitive impacts of untreated severe OSA, thereby highlighting the potential benefits of initiating CPAP therapy.

SUMMARY:
Objective: This observational, cross-sectional pilot study aims to assess "Brain Fog" (cognitive symptoms impacting memory, attention, and concentration) in severe Obstructive Sleep Apnea (OSA) patients. It compares two groups: those on CPAP treatment for at least 3 months and those not yet treated.

Procedures: Severe OSA patients (AHI > 30) will complete a 30-minute questionnaire at the Sleep Center Clinic, covering sociodemographic information, OSA diagnosis, and treatment details. Assessment scales will measure daytime sleepiness, sleep quality, and psychophysical fatigue.

Participants: 80 Sleep Center outpatients, evenly divided by age and gender:

40 with severe OSA on CPAP for at least 3 months. 40 with severe OSA not yet on CPAP. Duration: Approximately 12 months.

DETAILED DESCRIPTION:
This observational, cross-sectional, single-center pilot study aims to examine the presence of "Brain Fog" - a cluster of cognitive symptoms impairing memory, attention, and concentration - in patients with severe Obstructive Sleep Apnea Syndrome (OSA). It compares two groups: patients who have been undergoing CPAP treatment for at least 3 months and patients who have not yet begun treatment. Patients with severe OSA (AHI > 30), evaluated by a pulmonologist for CPAP therapy adaptation or already in therapy for at least 3 months, will be invited to participate in the study at the Sleep Center Clinic. After reviewing and signing informed consent, participants will receive a link to access the Qualtrics platform, where they will complete the online self-report questionnaire under the supervision of trained staff, available to assist if needed. The questionnaire, taking approximately 30 minutes to complete, will be administered once and will collect sociodemographic data (gender, age, marital status, educational level, occupational status, comorbidities, diagnosis date, CPAP adaptation start date, and COVID-19 health status over the past 12 months), including the Brain Fog Scale, currently undergoing Italian validation by our Research Group. Additional measures will include the Epworth Sleepiness Scale (ESS) to assess daytime sleepiness, the Pittsburgh Sleep Quality Index (PSQI) for sleep quality, the Fatigue Severity Scale (FSS), and Pichot's Fatigue Scale for psychophysical fatigue. The study anticipates recruiting 80 outpatients with severe OSA, evenly divided by age and gender into two groups: 40 patients on CPAP for at least 3 months and 40 patients who have not yet started CPAP. As no prior studies have investigated Brain Fog in OSA patients, conventional power calculations could not be applied; hence, 40 patients per group were deemed sufficient to provide preliminary estimates and identify any logistical or methodological issues for larger studies. Statistical analyses will be conducted using Jamovi 2.5.3 software, encompassing descriptive statistics, independent sample T-tests, Pearson's correlation to measure the strength of linear relationships between Brain Fog and other assessment scale scores, and a multiple regression model to examine the effect of independent variables on Brain Fog. In cases of non-normal data distribution, appropriate non-parametric analyses will be applied. The Brain Fog Scale, currently under Italian validation, may affect the reliability and validity of findings. Significant differences in Brain Fog levels are expected between CPAP-treated and untreated patients, with the hypothesis that treated patients will show symptom reduction. CPAP treatment is anticipated to improve memory, attention, concentration, and mental clarity in severe OSA patients. The collected data may also reveal a positive correlation between CPAP use, sleep quality improvement, and reduced Brain Fog symptoms. Furthermore, this study aims to provide preliminary data for calculating the necessary sample size for larger, more rigorous future studies. Clinical implications suggest that CPAP treatment may not only relieve respiratory symptoms of OSA but also offer significant benefits for cognitive functions, thus enhancing the quality of life for patients with severe OSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe OSA treated with CPAP for at least 3 months.
* Patients with severe OSA in new access and therefore not yet subjected to CPAP treatment.
* Patients with severe OSA who are able to understand the Italian language.

Exclusion Criteria:

* Patients who do not have a certified diagnosis of severe OSA.
* Patients with mild or moderate OSA.
* Patients with OSA who are unable to understand the Italian language.
* Patients with OSA who have neurological and/or oncological comorbidities, as verified by medical records.
* Patients with documented cognitive deficits, as verified by medical records.
* Patients with certified diagnoses of psychiatric disorders and/or substance use disorders (SUD), as verified by medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will be selected from a population of patients with severe Obstructive Sleep Apnea (OSA). Specifically, the population will include two distinct groups:
  Patients with Severe OSA Treated with CPAP: This group will consist of individuals who have been diagnosed with severe OSA and have been undergoing treatment with Continuous Positive Airway Pressure (CPAP) for at least three months. These patients are expected to have experienced a stabilization in their condition due to adherence to the CPAP therapy.
  Patients with Severe OSA in New Access: This group will include individuals who are newly diagnosed with severe OSA and have not yet started any treatment with CPAP. These patients will represent a baseline group to compare against those already receiving CPAP treatment.
  Both groups will consist of adult patients who are able to understand the Italian language, ensuring that they can accurately complete the self-report questionnaires involved in the study. Exclus
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Brain Fog | At enrollment only
  The Italian validation questionnaire is currently undergoing validation by our research group. In the original self-report scale, for each item, respondents are asked to indicate on a 5-point Likert scale (0 = "never", 1 = "rarely", 2 = "occasionally", 3 = "a lot of the time", 4 = "nearly all the time") how often they have experienced each symptom during the last two weeks. Total scale scores range from 0 to 92, with higher scores indicating increased levels of brain fog.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | At enrollment only
  self-report questionnaire designed to assess an individual's level of daytime sleepiness. It consists of eight questions that ask respondents to rate their likelihood of dozing off or falling asleep in various everyday situations, such as watching television, sitting in a car, or resting in the afternoon. Each item is scored on a scale from 0 to 3, where: 0 = Would never doze
  1. = Slight chance of dozing
  2. = Moderate chance of dozing
  3. = High chance of dozing The total score is calculated by summing the points from all eight questions, resulting in a possible score range from 0 to 24. Higher scores indicate greater levels of daytime sleepiness.
Pittsburgh Sleep Quality Index (PSQI) | At enrollment only
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized self-report questionnaire designed to assess sleep quality and disturbances over a one-month time period. It consists of 19 items that generate a global score based on seven component scores:
  Subjective Sleep Quality: Assesses the individual's perception of sleep quality.
  Sleep Latency: Measures the time taken to fall asleep. Sleep Duration: Evaluates the total amount of sleep obtained. Habitual Sleep Efficiency: Calculates the ratio of total sleep time to time spent in bed.
  Sleep Disturbances: Identifies problems that may disrupt sleep, such as waking up during the night.
  Use of Sleeping Medications: Assesses the frequency of sleep medication usage. Daytime Dysfunction: Evaluates the impact of sleep quality on daytime functioning.
  Each component is scored on a scale of 0 to 3, with higher scores indicating worse sleep quality. The global PSQI score ranges from 0 to 21, where a score greater than 5 is indicative of poor slee
Fatigue Severity Scale (FSS) | At enrollment only
  It is a self-report questionnaire designed to assess the severity of fatigue and its impact on daily functioning. It consists of nine statements related to fatigue, and respondents rate their level of agreement with each statement on a scale from 1 to 7, where:
  1. = Strongly Disagree
  2. = Disagree
  3. = Somewhat Disagree
  4. = Neutral
  5. = Somewhat Agree
  6. = Agree
  7. = Strongly Agree The statements focus on various aspects of fatigue, including how fatigue interferes with activities, its impact on motivation and physical performance, and the overall experience of fatigue in daily life. The total score is obtained by summing the ratings for all nine items, resulting in a possible score range from 9 to 63, with higher scores indicating greater fatigue severity.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Gnocchi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No
The data collection will also be conducted by Dr. Valentina Poletti, a member of my research group, who is pursuing her PhD on the same topic.

REFERENCES:
- [Result] Batool-Anwar S, Goodwin JL, Kushida CA, Walsh JA, Simon RD, Nichols DA, Quan SF. Impact of continuous positive airway pressure (CPAP) on quality of life in patients with obstructive sleep apnea (OSA). J Sleep Res. 2016 Dec;25(6):731-738. doi: 10.1111/jsr.12430. Epub 2016 May 30. PMID 27242272
- [Result] Rosenberg R, Thorpy MJ, Doghramji K, Morse AM. Brain fog in central disorders of hypersomnolence: a review. J Clin Sleep Med. 2024 Apr 1;20(4):643-651. doi: 10.5664/jcsm.11014. PMID 38217475
- [Result] McWhirter L, Smyth H, Hoeritzauer I, Couturier A, Stone J, Carson AJ. What is brain fog? J Neurol Neurosurg Psychiatry. 2023 Apr;94(4):321-325. doi: 10.1136/jnnp-2022-329683. Epub 2022 Dec 6. PMID 36600580